CLINICAL TRIAL: NCT03556787
Title: An Evaluation of a Gender Specific Insole to Provide Relief From Knee Pain Due to Osteoarthritis or General Anterior Knee Pain in Male Subjects When Used in Foot Wear Over a Period of Four Weeks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20244
Record Dates: First submitted 2018-06-04; First posted 2018-06-14 (Actual); Last update posted 2018-11-23 (Actual); Status verified 2018-11

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with knee pain (Experimental): Adults patients suffering from osteoarthritis pain or general knee pain
  Interventions: Device: BPI 1000013 (Dr Scholls Insole)

INTERVENTIONS:
Device: BPI 1000013 (Dr Scholls Insole) — Full length foam insole

SUMMARY:
The primary objective of this trial is to demonstrate the ability of a full length foam insole to provide relief from pain due to osteoarthritis of the knee or general knee pain when used in foot wear for a 4-week period of time.

The secondary objectives comprise the evaluation of the insole's ability to provide appropriate shoe fit and comfort as well as relief from osteoarthritis/ general knee pain after short-term use. The safety and tolerability of the test articles in terms of adverse events (AE) will also be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects with age 18 to 70 years and a self-reported foot size between 8 and 14
* Subjects with regular knee pain
* Subjects with a baseline pain level of pain of ≥20 mm to ≤90 mm on 100 mm VAS scale at baseline (Visit 1)
* Subjects must be able to walk unaided by cane or walker.

Exclusion Criteria:

* Subjects with knee pain which is due to a recent injury

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2018-06-04 (Actual); Primary Completion 2018-11-08 (Actual); Study Completion 2018-11-08 (Actual)

PRIMARY OUTCOMES:
Osteoarthritis knee pain according to Visual Analog Scale | Up to 4 weeks
  100 mm Visual Analog Scale: 0 = no pain to 100 = worst pain possible
General anterior knee pain according to Visual Analog Scale | Up to 4 weeks
  100 mm Visual Analog Scale: 0 = no pain to 100 = worst pain possible

SECONDARY OUTCOMES:
Foot Comfort according to Likert scale | Up to 4 weeks
  7-point Comfort/ Discomfort Likert scale, ranging from 1 = Extreme Discomfort to 7 = Extreme Comfort
Shoe Fit according to Likert scale | Up to 4 weeks
  7-point Comfort/ Discomfort Likert scale, ranging from -3 = Much too loose fit to 3 = Much too tight fit
Number of subjects with adverse events | Up to 4 weeks
Number of subjects with serious adverse events | Up to 4 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Focus & Testing, Inc., Calabasas, California
  - The Wolf Group, Cincinnati, Ohio